CLINICAL TRIAL: NCT05135195
Title: A Virtual Reality Platform Simulating Visual Impairment for Testing of Electronic Travel Aids and Performing Orientation and Mobility Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 21-00925
Record Dates: First submitted 2021-11-17; First posted 2021-11-26 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Visual Impairment; Age-Related Macular Degeneration; Diabetic Retinopathy; Glaucoma
MeSH Terms: conditions — Vision Disorders; Macular Degeneration; Diabetic Retinopathy; Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First Set of Experiments (Experimental): The anticipated number of participants is 336. All participants have healthy vision.
  Interventions: Other: In-House Developed VR Platform - AMD, DR, Glaucoma
- Second Set of Experiments (Experimental): The anticipated number of participants is 100. Of these, 80 participants have healthy vision, and 20 have glaucoma.
  Interventions: Other: In-House Developed VR Platform - Glaucoma

INTERVENTIONS:
Other: In-House Developed VR Platform - AMD, DR, Glaucoma — Participants will conduct experiments using commercial VR headsets and controllers. Visual impairments will be systematically simulated in VR. There are three visual impairment simulations (AMD, DR, and glaucoma) at three levels of severity (mild, moderate, or severe). Symptoms' simulation tools include a gaussian blur shader, distortion shader, and a culling mask with a gray spot in the middle.
  Arms: First Set of Experiments
Other: In-House Developed VR Platform - Glaucoma — In the second set of experiments, a multidimensional visual impairment simulation of a single pathology (glaucoma) will be used at three levels of severity (mild, moderate, or severe). The post-processing package to simulate includes glare, difficulty in light, change adaptation, ambient occlusion, visual clutter, and overall blurred effect. The shader graph package will be used to create a distortion localized on assets surfaces only.
  Arms: Second Set of Experiments

SUMMARY:
In this study, the study team utilize virtual reality (VR) to simulate visual impairments of different types and severity in healthy subjects. The platform implements three of the most widespread forms of visual impairment in the United States (US): age-related macular degeneration (AMD), diabetic retinopathy (DR), and glaucoma, each with three levels of severity, (mild, moderate, and severe). At present, glaucoma is further developed toward a multidimensional visual impairment simulation.

The platform is utilized: i) to provide a safe, controllable, and repeatable set of environments for development and preliminary testing of electronic travel aids (ETAs) in a variety of conditions (i.e., using the ETA to navigate in the immersed environment); and ii) to equip blind and low vision (BVI) professionals, inclusive of orientation and mobility (O&M) instructors, with a controlled, tunable training platform for skill/capacity building, assessment, and refinement of O&M techniques, as well as visually impaired trainees with a safe and immersive environment to improve their O&M skills and learn novel techniques. Two sets of hypothesis-driven experiments are proposed to assess the feasibility of the platform with respect to these two objectives.

ELIGIBILITY:
Inclusion Criteria (patients with visual impairment)

1. Aged 18-80;
2. People with glaucoma of all different levels and etiologies.

Inclusion Criteria (healthy controls)

1. Aged 18-80;
2. Gender neutral: male or female.

Exclusion Criteria (patients with visual impairment & healthy controls)

1. Significant cognitive dysfunction (score <24 on Folsteins' Mini Mental Status Examination)
2. Previous neurological illness or psychiatric disorders, or suffer from a heart condition or other serious medical conditions
3. Significant mobility restrictions; people using walkers and wheelchairs
4. Pregnancy
5. Elderly
6. Seizures (people who previously have had a seizure, loss of awareness, or other symptom linked to an epileptic condition)
7. Interference with medical devices (the headset and controller(s) may contain magnets or components that emit radio waves, which could affect the operation of nearby electronics, including cardiac pacemakers, hearing aids, and defibrillators)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2021-10-24 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Average time to complete the trial | 1 Day of Intervention
Average number of obstacle collisions during the trial | 1 Day of Intervention
Average travel time | 1 Day of Intervention
Average distance traveled by the participant | 1 Day of Intervention
Preferred walking speed | 1 Day of Intervention
Orientation | 1 Day of Intervention
  Orientation is measured through the time average of a polarization index, measured as the cosin of the angle between the direction of the instantaneous velocity vector and the straight line linking the instantaneous position of the participant and the following waypoint.
Number of instances in which the participant stop for more than 2 seconds | 1 Day of Intervention
Total time spent during stops of more than 2 seconds | 1 Day of Intervention
Average time it takes to understand how to interact with the system and run the simulation of the bus ride | 1 Day of Intervention

CONTACTS AND LOCATIONS:
Overall Officials: John-Ross Rizzo, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be available upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to Johnross.rizzo@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.